CLINICAL TRIAL: NCT00003136
Title: A Phase I/II Dose Escalation Trial of Carboplatin With Amifostine Pretreatment to Augment High Dose Cyclophosphamide With Autologous Peripheral Blood Stem Cell Support for the Treatment of Patients With Epithelial Ovarian Cancer
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Epithelial Ovarian Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8433; UCCRC-8433; ALZA-97-005-ii; NCI-V97-1357
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Amifostine; Carboplatin; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Cyclophosphamide (40mg/kg/day on days -6, -5 and -4), Carboplatin (1600, 1700 or 1800 mg/m2 on days -6, -5, -4 and -3), Amifostine (910 mg/m2 on days -6, -5, -4 and -3), Peripheral blood stem cell transplantation (day 0), G-CSF (beginning day 4)
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: carboplatin; Drug: cyclophosphamide; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: carboplatin
Drug: cyclophosphamide
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of amifostine, carboplatin and cyclophosphamide, followed by peripheral stem cell transplantation, in treating patients with epithelial ovarian cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of high dose carboplatin with a fixed dose of high dose cyclophosphamide with amifostine pretreatment, and peripheral blood stem cell rescue in patients with ovarian epithelial cancer. II. Monitor engraftment kinetics such as granulocyte and platelet recovery. III. Determine the toxic effects of this regimen in this patient population. IV. Document the response of this patient population to this regimen in terms of time to progression, event free survival, and overall survival.

OUTLINE: This is a dose escalation study. Patients undergo apheresis over 2-4 days to mobilize peripheral blood stem cells (PBSC). They then receive amifostine IV over 15 minutes. Fifteen minutes later, carboplatin is administered over 30 minutes on days -6 through -3. Cyclophosphamide IV is administered 1 hour after the carboplatin infusion is completed on days -6 through -4. PBSC are infused on day 0. Filgrastim (G-CSF) is administered beginning on day 4. Cohorts of 3-6 patients are treated at each dose level. At least 15 days must pass between the day of PBSC infusion and the next dose escalation. The dose limiting toxicity (DLT) is defined as the dose producing grade 3 or 4 nonhematologic toxicity in 2 of 6 patients. The maximum tolerated dose (MTD) is defined as one dose level below the DLT dose. At least 6 patients are treated at the MTD. Patients are followed monthly for 6 months, every 2-3 months for 1 year, and annually until death.

PROJECTED ACCRUAL: This study will accrue 28 patients over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven ovarian epithelial cancer or primary peritoneal carcinoma No tumors of low malignant potential Chemotherapy sensitive disease Relapse greater than 6 months after complete response to chemotherapy Partial response to most recent chemotherapy No more than 3 prior chemotherapy regimens Evidence of refractory or recurrent disease other than elevated CA-125 after primary surgery or chemotherapy; persistent disease need not be still present No brain metastases

PATIENT CHARACTERISTICS: Age: 65 and under Performance status: GOG 0 or 1 Life expectancy: Not specified Hematopoietic: WBC greater than 2500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal Renal: Creatinine clearance at least 50 mL/min Cardiovascular: Normal radionuclide cardiac scan with ejection fraction greater than 45% OR Normal left ventricular function by echocardiogram OR Cardiac clearance by Cardiology service Pulmonary: DLCO greater than 50% predicted Other: Not pregnant Hepatitis B and C negative HIV-1 negative

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1996-12; Primary Completion 2000-12 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David L. Grinblatt, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States